CLINICAL TRIAL: NCT07310719
Title: Selective Laser Trabeculoplasty Versus Latanoprost as First Line Treatments for Primary Open-angle Glaucoma and Ocular Hypertension: A Comparative Analysis
Brief Title: A Comparative Study of Intraocular Pressure Control Using Selective Laser Trabeculoplasty and Latanoprost as Initial Treatments for Primary Open Angle Glaucoma and Ocular Hypertension in Lagos State University Teaching Hospital
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lagos State Health Service Commission (Other)
Responsible Party: Principal Investigator, Anne Abang-Obi, Principal Investigator, Lagos State Health Service Commission
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LagosSHSC
Record Dates: First submitted 2025-12-09; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Primary Open Angle Glaucoma or Ocular Hypertension
Keywords: Selective laser trabeculoplasty
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Latanoprost 0.005% (Active Comparator): Latanoprost is an ocular hypotensive prostaglandin F2-alpha isopropyl ester prodrug that lowers IOP by increasing aqueous humour outflow through the uveoscleral pathway. Evidence from experimental and clinical trials suggests that Prostaglandin analogs are first-line agents as medical therapy for glaucoma because of the higher IOP-lowering effect, lower systemic side effects, and once daily dosing compared with other classes of drugs. Participants in this group will be required to instill latanoprost in both eyes daily in the evenings.
  Interventions: Other: Latanoprost (0.005%)
- Selective laser trabeculoplasty (Experimental): Selective laser trabeculoplasty is a non-invasive, laser-based treatment that targets specific cells in the trabecular meshwork (TM) to improve aqueous humor outflow, thereby reducing intraocular pressure in patients with glaucoma or ocular hypertension. The selective nature of SLT reduces collateral tissue damage, making it a more advantageous option compared to other laser treatments, as it preserves surrounding tissue while effectively targeting the trabecular meshwork
  Interventions: Procedure: Selective laser trabeculoplasty

INTERVENTIONS:
Procedure: Selective laser trabeculoplasty — Selective laser trabeculoplasty is a laser based treatment that reduces intraocular pressure. it is a safe alternative to medical therapy and surgery.
  Arms: Selective laser trabeculoplasty
Other: Latanoprost (0.005%) — Latanoprost is a prostaglandin analogue, a first-line ocular hypotensive medication because of it's high intraocular pressure lowering efficacy.
  Arms: Latanoprost 0.005%

SUMMARY:
The goal of this clinical trial is to compare the short-term efficacy and safety of selective laser trabeculoplasty (SLT) to 0.005% latanoprost eye drops in lowering intraocular pressure (IOP) as primary therapy in treatment-naïve patients diagnosed as early to moderate primary open-angle glaucoma(POAG) or ocular hypertension (OHT) in the Lagos State University Teaching Hospital, Ikeja. The main questions it aims to answer are:

1. Will Selective Laser Trabeculoplasty be an equally effective treatment option compared with 0.005% Latanoprost eyedrops in reducing Intraocular Pressure when used alone as first-line therapy in Nigerian patients with POAG and OHT?
2. Will Selective Laser Trabeculoplasty record a similar safety profile compared with 0.005% Latanoprost when used independently as a primary therapy?
3. How will the quality of life of patients who undergo Selective Laser Trabeculoplasty treatment compare with patients on 0.005% Latanoprost eyedrops?

Participants will be randomized to one of the two intervention groups. Group A(latanoprost group) will use 0.005% latanoprost eye drops every night at 2100hours(9.00pm) west African Time for 3 months. intraocular pressures will be monitored at intervals for a period of 3 months.

Group B(SLT group) will have Laser treatment administered as a one-off treatment. intraocular pressures will be monitored at intervals for a period of 3 months.

A record of side effects will be documented at each follow up visit

DETAILED DESCRIPTION:
STUDY AREA The research will be conducted at the Glaucoma clinic, Department of Ophthalmology, Lagos State University Hospital, Lagos, Nigeria. The hospital is one of the three tertiary centers in the state, delivering high-level healthcare services to the inhabitants of Lagos State and its surrounding communities. The Eye department's team includes consultant ophthalmologists, ophthalmic resident doctors, optometrists, ophthalmic nurses, pharmacists, medical record officers, account officers, and health attendants. The glaucoma clinic has a weekly throughput of approximately twenty new glaucoma patients and offers a comprehensive range of services, including optical, medical management, laser therapy, and surgical interventions. Patients are referred to the clinic from various sources, including the hospital's general outpatient department, as well as general and private hospitals within and outside Lagos state. There are two glaucoma clinic days in a week, and a total of approximately eighty-five glaucoma patients are seen per week with a staff strength of about seven.

STUDY DESIGN This is an observer-masked, prospective, randomized controlled trial. STUDY DURATION The study will be conducted over twelve months and will include data collection, analysis, results, and the conclusion of the thesis.

SAMPLE SIZE Total sample size for the study will be 138, 69 eyes per intervention group For this clinical analysis, the unit of analysis will be the eye. The sample size of eyes will be the available number of eyes from the number of patients recruited to the study.

ETHICAL CONSIDERATION The study will be submitted for ethical review and approval to the Lagos State University Teaching Hospital (LASUTH) Ethics and Research Committee. Written informed consent will be obtained from each participant following a detailed explanation of the study's purpose and procedures. Participant data will be kept confidential and the research will adhere to the tenets of the Helsinki Declaration

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18years and above.
2. Patients newly diagnosed as Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT).
3. Patients with elevated IOP greater than 21mmHg (average of 3 measurements taken on 3 different clinic visits).
4. Patients categorized as early or moderate glaucoma POAG (cup -disc ratio 0.5 to 0.7, visual field analysis MD - 6dB to -12dB and disc damage likelihood score (DDLS) 5 to 7) on funduscopy, Optical coherence tomography, and fundus photograph
5. Patients who agree to participate in the study after informed consent.

Exclusion Criteria:

1. A prior medical, surgical, or laser treatment for glaucoma
2. Patients diagnosed with primary congenital glaucoma or secondary glaucoma
3. Advanced glaucoma (CDR greater than 0.8, visual field analysis MD more than -12dB and DDLS stage 8 and above)
4. Patients with cloudy cornea or corneal opacity that would impair the view of the anterior chamber angles, fundus, or give false IOP readings
5. Patients with media opacity, such as cataracts, vitreous haze, or vitreous hemorrhage that prevents examination of the posterior segment.
6. Patients who have undergone previous ocular surgeries (cataract surgery, trabeculectomy).
7. Patients with a history of ocular trauma or uveitis
8. Pregnant and lactating women.

   -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Percentage intraocular pressure reduction from baseline | 3 months
  To compare the percentage reduction in IOP from baseline using SLT and 0.005% Latanoprost eye drops, each used independently as primary therapy over 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof B. Adekoya, FWACS, MD, Study Director — Lagos State University
Locations (1):
- Lagos State University teaching Hospital Eye Institute, Ikeja, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and study results
Supporting Information: Study Protocol, CSR
Time Frame: Requests for data can be submitted 9 months after article is published and data will be accessible for up to 3 years.
Access Criteria: Access to Individual Participant Data (IPD) may be requested by researchers carrying out Independent Scientific research after a research proposal, Statistical Analysis Plan (SAP) and Data Sharing Agreement (DSA) are reviewed, approved and signed.
URL: https://docs.google.com/file/d/1NDKJ_bd9rd3KeEcrl4O9WF2-9XG-GMFE/edit?usp=docslist_api&filetype=msword